CLINICAL TRIAL: NCT03641469
Title: Green Sun Medical Dynamic Scoliosis Brace
Acronym: GSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Sun medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.0
Record Dates: First submitted 2018-05-31; First posted 2018-08-22 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; thoracolumbosacral orthosis; spinal orthotic; health-related quality of life; treatment adherence
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Current TLSO users will crossover to use of the GSM brace.
Masking Description: The outcomes assessor will be blinded to brace type when measuring the out-of-brace x-ray.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Green Sun Dynamic Brace (Experimental): Historical measures of brace effectiveness (in- and out-of-brace Cobb angles), wear time, and brace-related quality of life will be compared to those measured after the subject is fit with a Green Sun dynamic brace.
  Interventions: Device: Green Sun Dynamic Brace

INTERVENTIONS:
Device: Green Sun Dynamic Brace — Change from standard-of-care TLSO to GSM brace

SUMMARY:
This is a pilot study to collect preliminary short-term data concerning the safety and performance of the Green Sun Dynamic brace in a sample of subjects with adolescent idiopathic scoliosis who are currently being treated with a TLSO.

DETAILED DESCRIPTION:
The Green Sun Medical Dynamic Brace (GSM) brace was developed as an alternative to rigid thoracolumbosacral orthoses (TLSOs, braces) commonly used to prevent continued curve progression in patients with adolescent idiopathic scoliosis (AIS). The brace applies corrective forces to the muscular and bony structures of the spine while preserving range of motion (ROM). The orthosis is prefabricated and adjusted for each patient. A series of semi-rigid segments encircle the patient's torso in close contact and are joined by a structure of flexible elements. These flexible (or elastic) elements generate stabilizing forces, providing the necessary immobilization while allowing relative motion of the semi-rigid segments. To date, this brace has been tested in the lab on healthy volunteers.

This study will recruit patients currently using a TLSO and compare the curve correction achieved in the GSM brace to that in their current brace. After 3 months in the GSM brace, the out-of-brace Cobb angle will be measured and compared to that at enrollment. Safety will be continually assessed. Brace-related quality of life (comfort, stress, interference with activities) will be self-reported. Adherence to the brace prescription will be measured using an in-brace temperature monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AIS
2. Current treatment with a TLSO, of ≥5 months' duration
3. Existing 3D surface scan of torso and out-of-brace x-ray within the past 6 months
4. One curve apex below T7
5. Ability to read and write English
6. Age 10-15 years
7. Female sex

Exclusion Criteria:

1) Parents/patients who decline participation and/or do not sign the consent/assent documents 2) Pregnant women 3) Unwilling or unable to return for follow-up visits

-

Ages: 10 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Haggard, Principal Investigator — Green Sun medical
Locations (7):
- United States (7):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Shriners Children's Southern California, Pasadena, California
  - Shriners Hospitals for Children - Northern California, Sacramento, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Shriners Children's St. Louis, St Louis, Missouri
  - National Scoliosis Center, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 patients with AIS were enrolled at 6 centers across the US. Recruitment opened May 2018 and continued until January 2024. Enrollment and study procedures were interrupted for several months by COVID in 2020.
Groups:
- Green Sun Dynamic Brace: TLSO at Baseline followed by GSM brace for 3 months
Period: Overall Study
Arm/Group | Green Sun Dynamic Brace
Started | 36
Completed | 25
Not Completed | 11
Not completed — Ineligible | 2
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Excluding 2 enrolled but ineligible subjects
Groups:
- Green Sun Dynamic Brace: Eligible subjects treated with a TLSO at baseline
Arm/Group | Green Sun Dynamic Brace
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 34
Out-of-brace Cobb angle at Baseline [Mean (Standard Deviation); unit: degrees] — Population: Baseline Cobb angle measurements (from x-ray taken within 180 days prior to baseline) not available for 6 subjects
  degrees
    number analyzed (Participants) | 28
    (all) | 30.68 (9.16)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Acceptable GSM In-Brace Correction
Description: Acceptable GSM in-brace correction was defined as a difference of 10 degrees or less between the TLSO and GSM in-brace Cobb angles.
Time Frame: Baseline (TLSO measurement) to GSM brace delivery (GSM measurement) within 60 days
Population: 24 subjects had x-rays in the TLSO and the GSM taken within a 60-day time frame.
Measure: Number; unit: Percentage acceptable GSM correction
Groups:
- Green Sun Dynamic Brace: Patients transitioned from current TLSO to GSM brace
Arm/Group | Green Sun Dynamic Brace
Number analyzed (Participants) | 24
Percentage acceptable GSM correction | 100

2. Primary Outcome: Percentage of Participants With Curve Stability or Progression at 3-month Follow-up
Description: Curve stability is defined as progression of 10 degrees or less between the Cobb angle at baseline and at follow-up after GSM wear (Baseline Cobb angle minus follow-up Cobb angle).
Time Frame: Baseline to ~3 mo Follow-up
Population: 28 patients had baseline out-of-brace x-rays taken within 6 months of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Green Sun Dynamic Brace
Number analyzed (Participants) | 20
Participants | 18

3. Primary Outcome: Unanticipated Adverse Events
Description: Unanticipated adverse events associated with the GSM brace and patient characteristics likely to raise safety issues
Time Frame: Up to 1 year
Measure: Number; unit: number of AE's reported
Arm/Group | Green Sun Dynamic Brace
Number analyzed (Participants) | 34
number of AE's reported | 1

4. Secondary Outcome: Change in Brace-related Quality of Life Scores (Brace Questionnaire)
Description: Change in Brace Questionnaire (BrQ) scores from baseline (reflecting experience with TLSO) to follow-up (reflecting experience with GSM brace). Total scores range from 20 to 100, with higher scores suggesting better quality-of-life during bracing. A positive change score suggests increased brace-related QOL related to exposure to the GSM brace.
Time Frame: Baseline to Visit 3 (3-4 months post-baseline)
Population: 14 subjects with both baseline and follow-up BrQ scores for analysis.
Measure: Median (Full Range); unit: Units on the scale
Arm/Group | Green Sun Dynamic Brace
Number analyzed (Participants) | 14
Units on the scale | 3.82 [-17.37 to 21.10]

5. Secondary Outcome: Change in Quality of Life Scores
Description: Change in scores on the Italian Spine Youth Quality of Life (ISYQOL) measure from baseline (reflecting experience with TLSO) to follow-up (reflecting experience with GSM brace). The total scores range from 0 to 100% where 100% indicates no problems related to spine or bracing issues. A positive change score suggests increased QOL related to exposure to the GSM brace.
Time Frame: Baseline to Visit 3 (3-4 months post-baseline)
Population: 12 subjects had baseline and follow-up ISYQOL scores for analysis
Measure: Median (Full Range); unit: change in percentage QOL
Arm/Group | Green Sun Dynamic Brace
Number analyzed (Participants) | 12
change in percentage QOL | 5.36 [-19.02 to 18.55]

6. Secondary Outcome: Difference in Vital Capacity Measured in TLSO and GSM Brace
Description: Lung vital capacity measured in the TLSO and in the GSM brace to estimate chest wall movement difference. Positive difference favors GSM.
Time Frame: Baseline
Population: Participants tested prior to March 2020, after which spirometry testing was stopped due to COVID
Measure: Mean (Standard Deviation); unit: milliliters
Groups:
- Green Sun Dynamic Brace: Measurements taken in the TLSO and the GSM brace.
Arm/Group | Green Sun Dynamic Brace
Number analyzed (Participants) | 16
milliliters | 82.81 (470.80)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Any untoward or unfavorable medical occurrence in a participant, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Teams were asked to continuously surveil for AE's during study visits and phone contacts; all AE's were to be reported using a standard case report form. AE's prior to switch to GSM brace at baseline were not recorded.
Groups:
- Green Sun Dynamic Brace: Use of the Green Sun Dynamic Brace
Arm/Group | Green Sun Dynamic Brace
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Green Sun Dynamic Brace (N=34)
Pressure point of skin related to device (Skin and subcutaneous tissue disorders) | 1 (1) — Subject reported skin irritation in the left axillary area while wearing the GSM brace. The brace was altered and the irritation was resolved without need for medical intervention. Classified as "mild", "expected", "related" to the device.

LIMITATIONS AND CAVEATS:
1. Enrollment and data collection was interrupted by COVID (e.g. spirometry testing was suspended)
2. Of the 11 subjects who did not complete the 30 day visit (>75 days of follow-up), 6 were among the first 10 subjects enrolled.The GSM brace underwent design and materials changes during the trial, especially during the evaluation of the first 10 subjects.
3. One study site shut down before all subjects had finished the protocol, resulting in missing data (n=2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements are not uniform across the sites. The most restrictive agreement states that the site PI and sponsor agree present results only together with the other clinical study sites unless specific written permission is obtained in advance from Sponsor up to 1 year post-completion. After that, the PI can publish/present independently if Sponsor is given the opportunity to review and comment prior to dissemination.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03641469/Prot_SAP_000.pdf